CLINICAL TRIAL: NCT06029699
Title: High Flow Nasal Cannula Versus Non Invasive Positive Pressure Ventilation in Reducing Reintubation in Mechanically Ventilated Patient
Brief Title: High Flow Nasal Cannula Versus Non Invasive Positive Pressure Ventilation in Reducing The Rate of Reintubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Osman Shehata Abdelkareem, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFNC vs NIPPV
Record Dates: First submitted 2023-08-25; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Failure; Re-intubation Rate
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: When the patient become weanable from mechanical ventilation, the subjects were extubated immediately and randomly divided into two groups, with one group receiving HFNC (called HFNC group), the other group receiving NIPPV (called NIPPV group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow nasal cannula group (Active Comparator): patients put on high flow nasal cannula after extubation
  Interventions: Device: high flow nasal cannula
- non invasive positive pressure ventilation group (Active Comparator): patients put on non invasive positive pressure ventilation group after extubation
  Interventions: Device: non invasive positive pressure ventilation

INTERVENTIONS:
Device: high flow nasal cannula — device are used for weaning patients after mechanical ventilation extubation
  Arms: high flow nasal cannula group
Device: non invasive positive pressure ventilation — device are used for weaning patients after mechanical ventilation extubation
  Arms: non invasive positive pressure ventilation group

SUMMARY:
This is study aim to compare between high flow nasal canula (HFNC) and non invasive positive pressure ventilation (NIPPV) in reducing the rate of reintubation in mechanically ventilated patient with successful weaning

DETAILED DESCRIPTION:
* High-flow nasal cannula (HFNC) oxygen therapy comprises an air/oxygen blender, an active humidifier, a single heated circuit, and a nasal cannula. It delivers adequately heated and humidified medical gas at up to 60 L/min of flow and is considered to have a number of physiological effects: reduction of anatomical dead space, positive end expiratory pressure ( PEEP ) effect, constant fraction of inspired oxygen, and good humidification
* Noninvasive positive-pressure ventilation is a safe and effective means of improving gas exchange in patients with many types of acute respiratory failure . for example, adding noninvasive ventilation to standard therapy decreased the need for endotracheal intubation...For patients assigned to noninvasive ventilation, the ventilator was connected with conventional tubing to a clear, full-face mask with an inflatable soft-cushion seal and a disposable foam spacer to reduce dead space .After the mask had been secured, pressure support was increased to achieve an exhaled tidal volume of 8 to 10 ml per kilogram, a respiratory rate of fewer than 25 breaths per minute, the disappearance of accessory muscle activity (as evaluated by palpation of the sternocleidomastoid muscle), and patient comfort
* The effects of high-flow nasal cannula (HFNC) on adult patients with acute respiratory failure (ARF) are controversial. The investigators aimed to further determine the effectiveness of HFNC in reducing the rate of endotracheal intubation in adult patients with ARF by comparison to noninvasive positive pressure ventilation (NIPPV)

ELIGIBILITY:
Inclusion Criteria:

* All patient suffer from acute respiratory failure and intubated for mechanical ventilation and then extubated for weaning
* Age >18 years old

Exclusion Criteria:

* In patients less than 18 years old
* Any contradiction in using HFNC as trauma or surgery or obstruction of nasopharynx
* Any contradiction in using NIPPV as facial trauma ..surgery ..deformity..or upper airway obstruction or upper gastrointestinal bleeding or high risk of aspiration

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
the need for re-intubation and weaning success which will be measured by arterial blood gas ( ABG ) | baseline

SECONDARY OUTCOMES:
Duration of using of HFNC or NIPPV | up to 30 days
Length of hospital stay measured by days | up to 30 days
In - hospital mortality measured by number of died cases | up to 30 days
Adverse events | up to 30 days
  Adverse events (occurrence of nosocomial pneumonia based on clinical and laboratory and radiological finding, need for MV measured by re-intubation rate)
Incidence of any possible complications associated with the use of HFNC and NIPPV | up to 30 days

REFERENCES:
- [Background] Nishimura M. High-flow nasal cannula oxygen therapy in adults. J Intensive Care. 2015 Mar 31;3(1):15. doi: 10.1186/s40560-015-0084-5. eCollection 2015. PMID 25866645
- [Background] Meyer TJ, Hill NS. Noninvasive positive pressure ventilation to treat respiratory failure. Ann Intern Med. 1994 May 1;120(9):760-70. doi: 10.7326/0003-4819-120-9-199405010-00008. PMID 8147550
- [Background] Ni YN, Luo J, Yu H, Liu D, Ni Z, Cheng J, Liang BM, Liang ZA. Can High-flow Nasal Cannula Reduce the Rate of Endotracheal Intubation in Adult Patients With Acute Respiratory Failure Compared With Conventional Oxygen Therapy and Noninvasive Positive Pressure Ventilation?: A Systematic Review and Meta-analysis. Chest. 2017 Apr;151(4):764-775. doi: 10.1016/j.chest.2017.01.004. Epub 2017 Jan 13. PMID 28089816
- [Background] Fang G, Wan Q, Tian Y, Jia W, Luo X, Yang T, Shi Y, Gu X, Xu S. [Comparative study on pros and cons of sequential high-flow nasal cannula and non-invasive positive pressure ventilation immediately following early extubated patients with severe respiratory failure due to acute exacerbations of chronic obstructive pulmonary disease]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2021 Oct;33(10):1215-1220. doi: 10.3760/cma.j.cn121430-20210623-00939. Chinese. PMID 34955131
- [Background] Gomez-Merino E, Sancho J, Marin J, Servera E, Blasco ML, Belda FJ, Castro C, Bach JR. Mechanical insufflation-exsufflation: pressure, volume, and flow relationships and the adequacy of the manufacturer's guidelines. Am J Phys Med Rehabil. 2002 Aug;81(8):579-83. doi: 10.1097/00002060-200208000-00004. PMID 12172066